CLINICAL TRIAL: NCT03965728
Title: Multiple Dose Escalation Study in a Randomized, Double-blind, Placebo-controlled Design to Investigate Safety, Tolerability, Pharmacokinetics, Drug-drug Interaction and Exploratory Pharmacodynamics of Multiple Oral Doses of BAY1830839 in Healthy Male Participants
Brief Title: Study to Investigate Safety, Tolerability, Pharmacokinetics, and Drug-drug Interaction of Multiple Oral Doses of BAY1830839 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 19401; 2019-000632-26 (EudraCT Number)
Record Dates: First submitted 2019-05-27; First posted 2019-05-29 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Midazolam; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY1830839 arm (Experimental): Period 1: Dose 1, Dose 2, Dose 3, Dose 4, Dose 5 and Dose 6, single dose. Period 2: Dose 1, Dose 2 and Dose 3, once daily over 10 days. Dose 4 and Dose 5, twice daily over 10 days. Dose 6, single dose on Day 1, three times daily (TID) for 9 days (Days 2-10).
  Interventions: Drug: BAY1830839; Drug: Midazolam; Drug: Methotrexate
- Placebo arm (Placebo Comparator): Placebo tablets matching BAY1830839
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1830839 — Tablet, oral.
  Arms: BAY1830839 arm
Drug: Placebo — Tablet, oral.
  Arms: Placebo arm
Drug: Midazolam — For all dose steps. Oral. Two single doses. One dose administered during pre-dose in Period 1 and the second dose administered on the last day of treatment with BAY1830839 or placebo in Period 2
  Arms: BAY1830839 arm
Drug: Methotrexate — Only for Dose 3 step. Tablet, oral. Two single doses. One dose administered during pre-dose in Period 1 and the second dose administered on the last day of treatment with BAY1830839 or placebo in Period 2.
  Arms: BAY1830839 arm

SUMMARY:
The aim of this study is to investigate safety, tolerability and pharmacokinetics of increasing repeated oral doses of BAY1830839 in healthy male participants including the investigation of any potential drug-drug interactions of BAY1830839 with midazolam and methotrexate. In addition, the effects of BAY180839 on exploratory pharmacodynamics biomarkers in healthy participants will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Overtly healthy as determined by medical evaluation including (medical and surgical history, physical examination, laboratory tests, ECG, vital signs).
* Confirmation of the participant's health insurance coverage prior to the first screening examination/visit.
* Body Mass Index (BMI): above or equal 18.5 and below or equal 30.0 kg/m² at screening
* Male
* Study participants of reproductive potential must agree to utilize two reliable and acceptable methods of contraception simultaneously when sexually active. This applies for the time period between admission to the study site until 12 weeks after the last administration of the study intervention. The following contraceptive methods will be regarded as adequate in the context of this study:

condoms (male or female) with or without a spermicidal agent;

* diaphragm or cervical cap with spermicide;
* intra-uterine device;
* hormone-based contraception.

  * Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
  * The informed consent must be signed before any study specific tests or procedures are done.
  * Ability to understand and follow study-related instructions

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal.
* Relevant diseases within the last 4 weeks prior to the first study administration of study intervention.
* Febrile illness within 4 weeks before the first study administration of study intervention.
* Known hypersensitivity to any study intervention (active substances or excipients of the preparations) to be used in the study.
* Known severe allergies, significant non-allergic drug reactions, or multiple drug allergies, e.g. allergies to more than 3 allergens, allergies affecting the lower respiratory tract - allergic asthma, allergies requiring therapy with corticosteroids, or urticaria.
* Use of systemic or topical medicines or substances which oppose the study objectives or which might influence them within 4 weeks before first study drug administration, e.g. an investigational drug; any drug known to induce liver enzymes (e.g. dexamethasone, barbiturates, rifampicin, anticonvulsants, griseofulvin, St. John's Wort [Hypericum perforatum]).
* History of COVID-19 as patients with a history of severe COVID-19 infection.
* Incomplete SARS-CoV-2 vaccination

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Frequency of TEAEs | 7 days (period 1)
  TEAE: treatment-emergent adverse event
Frequency of TEAEs | 18 days (period 2)
Severity of TEAEs | 7 days (period 1)
Severity of TEAEs | 18 days (period 2)
AUC(0-24)md of BAY1830839 (QD and TID dosing) | Day 1 period 1
  QD:once daily administration TID: three times daily administration
AUC(0-12)md of BAY1830839 (BID dosing only) | Day 1 period 2
  BID:twice daily administration
Cmax,md of BAY1830839 after multiple dosing | 18 days (period 2)
Cav of BAY1830839 after multiple dosing | 18 days (period 2)
AUC of midazolam in plasma in presence/absence of BAY1830839 | Day -1 period 1
  If AUC(tlast-∞) >20% of AUC then AUC(0-tlast) will replace AUC.
Cmax of midazolam in plasma in presence/absence of BAY1830839 | Day -1 period 1
AUC of methotrexate in plasma in presence/absence of BAY1830839 | Day -1 period 1 (Dose group 3 of BAY1830839 only)
  If AUC(tlast-∞) >20% of AUC then AUC(0-tlast) will replace AUC.
Cmax of methotrexate in plasma in presence/absence of BAY1830839 | Day -1 period 1 (Dose group 3 of BAY1830839 only)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/